CLINICAL TRIAL: NCT04882865
Title: Apparatus and Method for Moving Patients: Users Impressions of the Use of a Novel Device to Assist With Patient Movement as Compared to Repositioning Sheets
Brief Title: Apparatus and Method for Moving Patients
Acronym: AMMP
Status: Active, not recruiting | Type: Observational
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: 30760
Record Dates: First submitted 2021-05-04; First posted 2021-05-12 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Respiratory Failure; Covid19
Keywords: prone ventilation; patient movement
MeSH Terms: conditions — Respiratory Insufficiency; COVID-19 | interventions — Insemination, Artificial, Heterologous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- healthy volunteers as "patients": use of the device (AMMP) and the process on 5 healthy volunteers undergoing proning, as well as "general care" (movement up or down the bed, rotated laterally). As well, repositioning sheets will be used for general care. Surveys of the impressions of team members of the value (ease of use, efficiency, safety, physical demands) of using the AMMP and the repositioning sheets with these "patients" will be completed.
  The impressions of the volunteers as patients will be surveyed, with particular reference to comfort and security during movement
  Interventions: Device: assist
- ICU patients severe respiratory failure: patients with severe respiratory failure eligible for prone ventilation will be recruited with surveys provided to team members to gauge their impressions of the value of using the AMMP with the proning process for these patients. Surveys for 40 proning processes will be obtained. Movement from back to stomach or from stomach to back is considered a single process. A single patient may undergo multiple proning processes as prone ventilation is delivered for several days, with multiple healthcare team members participating in their care. We anticipate this will involve 10 patients, and 3 team members to be involved with each proning process.
  Interventions: Device: assist
- Patients admitted to the ICU: 40 patients will have the AMMP used for general care. An additional 40 will have repositioning sheets used for general care. Healthcare team members involved with the care of these patients will be surveyed re their impressions of the value of using the AMMP or the repositioning sheets. We cannot predict the number of healthcare team members involved with the care of each patient s because of clinical conditions and length of stay
  Interventions: Device: assist

INTERVENTIONS:
Device: assist — A custom designed patient wrap will envelope the patient. This will be coupled to a mechanical lift system to facilitate repositioning of the patient (AMMP) Commercially available repositioning sheets will be used for the general care of some study patients

SUMMARY:
A novel device and process to move patients has been developed, particularly useful for patients with severe respiratory failure (ie COVID 19) who require prone ventilation (moving from their back onto the stomach and then onto back for a 16 hour cycle, usually for several days).

This study will assess staff impressions of the feasibility of the use of this device/ process to prone patients as well as their impressions of the use of this device, compared to repositioning sheets, for the general care of the ICU patient. An economic analysis of the use of the AMMP for proning compared to movement without assists will be done

DETAILED DESCRIPTION:
Movement of non ambulatory patients is typically a physically demanding, resource intensive intervention that places the healthcare team members at risk of injury. A quantitative survey of healthcare team members perspectives on the challenges associated with patient movement will be distributed.

This is particularly true for caregivers responsible for severely ill respiratory failure patients (ie COVID 19) who are moved into prone position (flipped on to their stomach) and back to supine over a 16 hour cycle, typically repeated for several days, as part of their therapy. (proning) A method of wrapping the patient in a secure "cocoon" which is coupled to a mechanical lift system through a designed strapping system and support bar will be tested for proning on healthy volunteers and then in the clinical environment ( intensive care unit (ICU) . Healthcare team members will complete surveys to assess ease of use, efficiency, safety and physical demands of this process relative to traditional (control) manual methods of patient reorientation, without the use of assists for proning.

Critically ill nonambulatory patients require assistance to move. The AMMP can be used to assist and impressions of this device. Comparing the impressions of healthcare team members of the use of the AMMP, repositioning sheets, and to care without the use of a movement assistance device will be undertaken using quantitative surveys An economic analysis of the use of the AMMP to prone patients, focused on personnel time and personal protective equipment use, compared to proning without assistance, will be completed

ELIGIBILITY:
Inclusion Criteria:any adult ICU patient is eligible for enrolment in assessment of health care team members impressions of the use of repositioning sheets for general care ( movement up or down the bed or in to lateral position) Adult ICU patients admitted to the ICU with severe respiratory failure (PaO2/FiO2 ratio <150) are candidates for use of the AMMP for prone positioning unless exclusion criteria are present Adult ICU patients requiring general care are candidates for use of the AMMP for general care unless exclusion criteria are present -

Exclusion Criteria:discretion of ICU attending, unable to obtain consent, unstable spine fracture, chest tube drainage in place, open abdomen, >140 kg

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: adult (>16y) patients admitted to the Med- Surg Neuro ICU at the Queen Elizabeth II Health Science Centre, including those with severe respiratory failure.
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Perception of the experience of "healthy volunteers as patients" when moved by a healthcare team utilizing a novel device (AMMP) or repositioning sheets. | 6 months to 12 months
  The AMMP will be used to move volunteers for "general care" (up or down the bed, into lateral position) or into prone position. The repositioning sheets will be used to move volunteers for "general care". Repositioning sheets are not designed to be used for prone positioning Qualitiative surveys of the "patient" experience utilizing a survey tool with a 5 point Likert scale will be used focused on their perceptions of comfort, anxiety related to the movement and feelings of feeling security as well as open narrative
Perception of healthcare team members of the use of repositioning sheets and the AMMP to assist with patient handling of ICU patients requiring general care ( movement up or down the bed, into lateral position) | 6 months to 12 months
  Repositioning sheets and the AMMP will be used by healthcare team members to facilitate patient handling for general care of ICU patient in an ICU where this type of movement aid has not been previously utilized. Qualitiative review of team members impressions of the feasibility of the use of this device for this purpose will be assessed utilizing surveys with 5 point Likert scale as well as open narrative. Team members impressions of the use of this aid, compared to the AMMP for general care and to their impressions of the provision of general care without the use of aids will be assessed in the survey tool
Perception of healthcare team members of the use of a novel process to assist with patient handling in the ICU, in particular for movement into prone position | 6 months to 12 months
  A novel apparatus and method to reposition patients ( AMMP) has been developed. Perceptions of team members using this to move ICU patients from supine to prone, or prone to supine, during therapy for severe respiratory failure, will be assessed relative to traditional approaches to movement of patients without aids. A quantitative analysis of perceptions across multiple dimensions (ease of use of the device, efficiency, physical demand for healthcare team member, adverse effects on patients) will be undertaken utilizing a survey instrument with a 5 point Likert scale as well as open narrative

SECONDARY OUTCOMES:
Economic analysis of the use of the AMMP for ICU patients requiring prone ventilation | 6-12 months
  Movement of patients from supine to prone or prone to supine to facilitate mechanical ventilation for patients with severe lung disease is resource intensive (requirement for personal protective equipment (PPE)) , dependant on a large team (5-7 people) and time intensive. A comparison of the efficiency of patient movement with the AMMP relative to movement without an aid will be completed. Historical values for time to complete, number of personnel needed to complete and the number of sets of PPE for this process will be compared to these parameters when the AMMP is used. Personnel costs (number of people x cost per hour x total time taken) and resource utilization ( number of sets of PPE x cost /set of PPE) added together will define "total costs" for this comparison

OTHER OUTCOMES:
perceptions of healthcare tram members of difficulties in handling patients | 3 months
  Non ambulatory patients must move, or be moved, to recover. Healthcare team members frequently must assist, which is physically demanding, putting team members at risk of injury. The concerns of healthcare team members in the acute care ( ICU) will be surveyed to collate and quantify their role in the healthcare team, their experience with patient handling, opinions on ideal team size for patient handling, and injury history associated with patient handling

CONTACTS AND LOCATIONS:
Locations (1):
- Qe Ii Hsc, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No